CLINICAL TRIAL: NCT06823960
Title: An Italian Multicenter Retrospective Observational Study to Assess Effectiveness and Safety of Zanubrutinib for Patients With Marginal Zone Lymphoma Treated in Italy Under the Named Patient Program (NPP)
Brief Title: Study to Assess Effectiveness and Safety of Zanubrutinib for Patients With Marginal Zone Lymphoma Treated in Italy Under the Named Patient Program (NPP)
Acronym: ZanOs
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ZanOs
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Marginal Zone Lymphoma(MZL)
Keywords: zanubrutinib
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational, non-interventional, retrospective, multicentre study focusing on efficacy and safety of zanubrutinib in daily clinical practice in patients with relapsed/refractory (R/R) marginal zone lymphoma.

DETAILED DESCRIPTION:
Due to the rarity of the condition and the novelty of its application, the study is intended to be exploratory, with the aim of providing interim evidence on which to plan future studies in larger populations. Data will be collected from the start of therapy until 6 months after the end of therapy, when applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of relapsed/refractory marginal zone lymphoma
2. Patients who received at least one dose of zanubrutinib under the Named patient program (D.M. 7 Sep 2017), between January 2021 and October 2023 3) Age≥18 at start of zanubrutinib therapy. 4) Signature of written informed consent to study participation and personal data processing.

Exclusion Criteria:

1) relapsed/refractory marginal zone lymphoma patients who received zanubrutinib in a clinical trial context.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed/refractory marginal zone lymphoma treated with at least one dose of zanubrutinib under the Named patient program (D.M. 7 Sep 2017), between January 2021 and October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | through the duration of study, an average of 6 months
  the sum of the Complete Response [CR] and Partial Response [PR]) in accordance with the Lugano Classification

SECONDARY OUTCOMES:
Duration of response (DoR) | through the duration of study, an average of 6 months
  To evaluate safety and tollerability of zanubrutinib in patients with relapsed/refractory marginal zone lymphoma treated with at least one dose of zanubrutinib under Named patient program
Progression Free Survival (PFS) | through the duration of study, an average of 6 months
  To evaluate safety and tollerability of zanubrutinib in patients with relapsed/refractory marginal zone lymphoma treated with at least one dose of zanubrutinib under Named patient program
Overall Survival (OS) | through the duration of study, an average of 6 months
  To evaluate safety and tollerability of zanubrutinib in patients with relapsed/refractory marginal zone lymphoma treated with at least one dose of zanubrutinib under Named patient program
Best response rate (BRR), | through the duration of study, an average of 6 months
  To evaluate safety and tollerability of zanubrutinib in patients with relapsed/refractory marginal zone lymphoma treated with at least one dose of zanubrutinib under Named patient program
Disease Free Survival (DFS) | through the duration of study, an average of 6 months
  To evaluate safety and tollerability of zanubrutinib in patients with relapsed/refractory marginal zone lymphoma treated with at least one dose of zanubrutinib under Named patient program
Type, incidence, severity of any adverse events (AE) | from start of treatment to 30 days after last dose
  To evaluate safety and tollerability of zanubrutinib in patients with relapsed/refractory marginal zone lymphoma treated with at least one dose of zanubrutinib under Named patient program

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (15):
- Italy (15):
  - AOU SS Antonio e Biagio e Cesare Arrigo, Alessandria, Alessandria
  - IRCCS-AOU di Bologna, Bologna, Bologna
  - P.O. Garibaldi-Nesima_UOC Ematologia, Catania, Catania
  - AO di Cosenza, P.O. "Annunziata" - UOC di Ematologia, Cosenza, Cosenza
  - AOU di Ferrara_ UO di Ematologia - Dipartimento di Oncologia e Medicine Specialistiche, Ferrara, Ferrara
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST IRCCS, Meldola, Forlì Cesena
  - Istituto Clinico Humanitas IRCCS - UO Ematologia, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda _ UOC Ematologia, Milan, MIlano
  - IOV - Istituto Oncologico Veneto - IRCCS _UOC Oncologia1, Padua, Padova
  - Ospedali Riuniti Villa Sofia - Cervello _ UO di Ematologia ad Indirizzo Oncologico, Palermo, Palermo
  - Ospedale Santa Maria delle Croci- OU Ematologia di Ravenna, Ravenna, Ravenna
  - Fondazione PTV Policlinico Tor Vergata- U.O.C. Patologie Linfoproliferative, Roma, Roma
  - AOU Città della Salute e della Scienza, "Le Molinette" - Divisione di Ematologia, Torino, Torino
  - Ospedale Ca' Foncello, Azienda ULSS n. 2 Marca trevigiana - UOC Ematologia Dipartimento di Medicina, Treviso, Treviso
  - Azienda sanitaria universitaria Giuliano Isontina (ASU GI) - Ospedale Maggiore- SC (UCO) Ematologia, Trieste, Trieste

IPD SHARING:
Plan to Share IPD: No